CLINICAL TRIAL: NCT01520155
Title: CArdiovascular Risk Assessment STudy in Lupus Erythemathodes (CASTLE): Studie Zur Detektion Des kardiovaskulären Risikos in Patienten Mit Systemischem Lupus Erythematodes
Brief Title: CArdiovascular Risk Assessment STudy in Lupus Erythemathodes (CASTLE)
Acronym: CASTLE
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Fox, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: sleffm001
Record Dates: First submitted 2011-12-12; First posted 2012-01-27 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus erythematosus; cardiovascular risk
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Every participant will provide 20 ml Serum for further laboratory analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Systemic lupus erythematosus with renal affection: 30 patients will be investigated suffering from a known systemic lupus erythematosus with renal affection
- Systemic lupus erythematosus without renal affection: 30 patients will be investigated suffering from a known systemic lupus erythematosus without renal affection
- Non-autoimmune kidney disease: Patients with non-systemic, non-autoimmune kidney disease

SUMMARY:
The key of this prospective study is to identify a potentially increased cardiovascular risk in patients with systemic Lupus erythematodes, with and without renal affection. Three groups of patients will be compared.

DETAILED DESCRIPTION:
Key of this prospective study is to identify a potentially increased cardiovascular risk in patients with systemic Lupus erythematodes, with and without renal affection. Three group of patients will be compared as followed. First group are patients with known systemic Lupus erythematodes without renal affection, second group are patients with known systemic Lupus erythematodes with renal affection and the third group are patients with a non-autoimmun chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic Lupus erythematosus

Exclusion Criteria:

* Patients without systemic Lupus erythematosus

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without systemic Lupus erythematosus
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Identification of cardiovascular risk in patients with systemic Lupus Erythematodes | one year
  Identification of cardiovascular risk in patients with systemic Lupus Erythematodes

CONTACTS AND LOCATIONS:
Overall Officials: Joachim R Ehrlich, MD, Study Chair — Frankfurt University Academic Medical Center
Locations (1):
- Frankfurt University Academic Medical Center, Frankfurt am Main, Hesse, Germany